CLINICAL TRIAL: NCT06191198
Title: Communication Bridge: Optimizing an Evidence-based Intervention for Individuals With Primary Progressive Aphasia
Brief Title: Communication Bridge 3 Study
Acronym: CB3
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Western University, Canada (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB23-1175; 7R01AG055425-07 (NIH)
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Primary Progressive Aphasia
Keywords: Aphasia; Dementia; Communication; Frontotemporal Dementia; Alzheimer Disease
MeSH Terms: conditions — Aphasia, Primary Progressive; Aphasia; Dementia; Communication; Frontotemporal Dementia; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: NIH Stage 2 behavioral clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Communication Bridge™ (Experimental): Participants receive Communication Bridge™, a multi-component, participation-focused, dyadic intervention in which both the person with PPA and their co-enrolled communication partner are intervention recipients. Communication Bridge™ is modelled on the Living with Aphasia: Framework for Outcome Measurement (A-FROM) and the Care Pathway Model that was developed for persons living with primary progressive aphasia. Consistent with participation-focused intervention models personally salient training stimuli are incorporated into all therapy activities in the Experimental arm.
  Interventions: Behavioral: Communication Bridge™
- Evidence-Based Impairment Focused (Active Comparator): The Control arm includes a non-dyadic intervention in which the person with PPA is the active intervention recipient and their communication partner is in a supporting role. In the Control arm, participants receive a speech-language intervention designed to address impairment and functional limitations, comprised of activities that address word retrieval and 'automatic' speech production using fixed, non-personalized, stimuli across participants.
  Interventions: Behavioral: Evidence-Based Impairment Focused

INTERVENTIONS:
Behavioral: Communication Bridge™ — Evidence-based speech language therapy treatment will be compared and contrasted in the two arms of the study.
  Arms: Communication Bridge™
Behavioral: Evidence-Based Impairment Focused — Evidence-based speech language therapy treatment will be compared and contrasted in the two arms of the study.
  Arms: Evidence-Based Impairment Focused

SUMMARY:
This study will use a randomized controlled trial design to evaluate the effect of two evidence-based treatments for adults with mild-moderate Primary Progressive Aphasia (PPA). The aim of the study is to help us better understand the effects of speech-language therapy on communication abilities in individuals with PPA.

DETAILED DESCRIPTION:
Participants with a diagnosis of PPA and their actively-engaged care partners will be involved in the study for approximately 17 months. Each participant will receive a laptop equipped with the necessary applications and features for the study. Participants will receive up to 10 evaluations and 20 speech therapy sessions with a licensed speech therapist, as well as access to Communication Bridge, a personalized web application to practice home exercises that reinforce treatment strategies. There are no costs to participate in this study.

ELIGIBILITY:
Inclusion Criteria (person with PPA):

1. Meets diagnostic criteria for PPA based on neurologist and supporting medical assessments (extracted from medical records)
2. English as primary language used in daily communication activities (by self-report)
3. Adequate hearing (aided or unaided) for communicating with others in a crowded room (by self-report)
4. Adequate vision (aided or unaided) for reading a newspaper, or other functional materials (by self-report)
5. Able to pass technology screening and demonstrates sufficient knowledge for use of video conference and Communication Bridge™ web application use (with or without training)
6. Geriatric Depression Scale score ≤ 9
7. Mild-moderate PPA informed by a structured interview with a speech-language pathologist and a standardized testing battery.

Inclusion Criteria (Co-enrolled communication partner):

1. 18+ years of age
2. English as primary language used in daily communication activities (by self-report)
3. Adequate hearing (aided or unaided) for communicating with others in a crowded room (by self-report)
4. Able to pass technology screening* and demonstrates sufficient knowledge for use of video conference and Communication Bridge™ web application use (with or without training)

Exclusion Criteria:

* A dementia diagnosis other than Primary Progressive Aphasia
* Participation is co-enrolled in an outside speech language therapy program during the study course.
* Communication partners will be excluded if they have a pre-existing communication impairment that would affect study participation (e.g., aphasia, dementia)

Medical records will be requested and reviewed to determine eligibility

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2028-07-15 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in Communication Participation Person Centered Goals | 5 assessment time points through study completion (up to 18 months)
  Goal Attainment Scaling, a 7-point rating scale with -3 representing 'no longer participating' and +3 representing 'exceeded goal'. Higher scores indicate better progress in goal achievement.
Change in Communication Participation | 5 assessment time points through study completion (up to 18 months)
  The CPIB measure is a 10-item, disorder-generic, Likert scale that asks persons to rate how their condition interferes with participating in daily communication activities (e.g., talking to people you know/do not know, securing a turn in a fast-moving conversation). The psychometric properties of the measure have been published previously (Baylor et al., 2013; Baylor et al., 2019). Both raw and T-scores are available. The CPIB T-score has a theoretical mean of 50 and standard deviation of 10 with higher numbers reflecting higher levels of participation in communication activities.
Montgomery Burden Inventory (MBI) | 5 assessment time points through study completion (up to 18 months)
  The MBI is a pen/paper Likert scale with 16 items distributed across three subscales (Montgomery et al., 1985) completed by the care partner. Total and mean item scores are calculated for each of the three subscales: Objective burden is defined as the perceived infringement of disruption of tangible aspects of a caregiver's life; Subjective demand/relational burden is typically described as the extent to which the caregiver perceives that the care recipient is overly demanding in the context of caregiving; Subjective stress burden is the emotional impact of caregiving responsibilities. Participants rate each item with a score between 1 (Not at all) and 5 (A great deal) corresponding to the amount of perceived burden. Higher scores reflect increased burden. Internal consistency .81 to .90. Construct validity demonstrated in mixed cohort of care partners of persons with dementia. Test-retest stability coefficients are robust (ICC of 0.92 to 0.91) (Farley et al., 2010).

CONTACTS AND LOCATIONS:
Overall Officials: Emily Roglaski, PhD, Principal Investigator — Professor of Neurology
Locations (1):
- University of Chicago - American School Building, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes